CLINICAL TRIAL: NCT05050552
Title: Oxygen Reserve Index and Its Relations With Primary Hemodynamical and Oximeter Parameters During Elective Thoracic Surgical Operations
Brief Title: Oxygen Reserve Index in One-Lung Ventilation During Elective Thoracic Operations
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Dr Gonul Sagiroglu, Associate Professor of Anesthesiology and Reanimation, Trakya University
Other Study IDs: TrakyaH
Record Dates: First submitted 2021-09-06; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: One-Lung Ventilation; Hypoxemia During Surgery; Oxygen Reserve Index; Perfusion Index; Pleth Variability Index
Keywords: ventilation; hypoxemia; one-lung ventilation; oxygen; perfusion
MeSH Terms: conditions — Respiratory Aspiration; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Masimo Radical-7 Pulse CO-Oximeter — The Masimo Radical-7 Pulse CO-Oximeter is a device for the measurement of pulse oximetry, oxygen reserve index (ORi), perfusion index (PI), and pleth variability index (PVI). The device is the product of a company called Masimo Inc, Irvine, CA, USA

SUMMARY:
The investigators' goal is to perform an observational cohort study investigating the use of oxygen reserve index (ORi) in patients undergoing elective thoracic surgery and one-lung ventilation (OLV). For this purpose, ORi values are recorded and compared to the other collected hemodynamical and oximeter parameters. The primary hemodynamic parameters include heart rate (HR) and blood pressure (BP), while; oximeter device-related parameters include peripheral oxygen saturation, perfusion index (PI), and pleth variability index (PVI).

The investigators' secondary goal is to investigate relationships between these hemodynamical and oximeter parameters using statistical analysis methods.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the possible benefits of using the oxygen reserve index (ORi) parameter during one-lung ventilation (OLV) and elective thoracic operations. For this purpose, ORi values are compared to primary hemodynamical parameters of blood pressure (BP) and heart rate (HR) and Meanwhile, a device from Masimo Inc, USA, provides oximeter-related parameters, including peripheral oxygen saturation, perfusion index (PI), and pleth variability index (PVI). The secondary objective is to investigate possible statistically significant correlations between these hemodynamical and oximeter parameters using appropriate statistical methods.

The study participants are patients undergoing video-assisted thoracotomy surgical procedures (VATS) or open thoracotomy for suspicion and possible lung tumor removal. The surgical operation of either lobectomy, pneumonectomy, lung biopsy, or wedge resection is considered during this procedure. The inclusion and exclusion criteria are summarized in another section of the clinicaltrials.gov registration document. All patients in the study receive a similar anesthetic management protocol. Premedication is not required in the study. After admitting a patient to the operating theatre, pulse oximetry SpO2, electrocardiogram, and noninvasive blood pressure monitoring are established. Heart rate (HR), mean arterial pressure (MAP), systolic blood pressure (SBP), and diastolic blood pressure (DBP) are measured at certain time points. Anesthesia requires induction of anesthesia with intravenous doses of propofol (Pofol, Fresenius Pharmaceutical, Turkey), 2 to 3 mg/kg, rocuronium (Esmeron, Organon Pharmaceuticals, U.S.A.) at a dose of 0.6 mg/kg, and fentanyl (Janssen fentanyl, Janssen Pharmaceutical, Belgium) at a dose of 2 to 3 mcg/kg. Tracheal intubation requires the use of a left Robertshaw double-lumen tube. During anesthesia, one-lung ventilation (OLV) is provided to all patients in addition to mechanical ventilation. The anesthesia maintenance includes inhalational anesthetic of sevoflurane (Sevorane, Abbott Pharmaceutical, USA) at an end-tidal concentration of 1 to 2% to provide a sufficient minimum alveolar concentration to establish anesthesia and intravenous fentanyl boluses at a dose of 0.2 mcg/kg every hourly to provide analgesia and to keep mean arterial blood pressure between 60 and 80 mmHg. In addition to standard follow-up parameters, oxygen reserve index (ORi), perfusion index (PI), pleth variability index (PVI) is monitored for each patient at certain time points. Hypoxemia during OLV was defined as peripheral oxygen saturation (SpO2) value of less than 95% when the inspired oxygen fraction (FiO2)value is equal to or greater than 60% on a pulse oximetry device. Hemodynamic and oximeter data were continuously monitored. The parameters that are in need of investigation include; MAP, SBP, DBP, HR, SpO2, PaO2, ORi, PI, and PVI values. These data are monitored at thirteen different time points during the period of anesthesia induction and maintenance of the surgery. The device used in this study is called the Radical-7 Pulse CO-Oximeter device for the measurement of ORi, PI, and PVI. A correlation between these values was investigated on the continuous graphs. The duration of surgery, anesthesia, OLV, and total 100% oxygen application time are recorded. Blood gas analysis was provided at DL5 at a 5-minute time point and blood gas analysis was performed for prolonged surgeries and for surgeries with high bleeding performance that required other analysis. Routinely, patients are ventilated with 50% FiO2 (50% oxygen + 50% air mixture, 1 liter/minute fresh gas flow) after induction. The value of FiO2 rises depending on pulse oximeter values between the values of 60% and 100% in order to keep SpO2 values greater than 94. The incidence of thromboembolic complications, arrhythmia, pneumonia, the duration of hospital and intensive care unit stay is recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients at ages between 22 to 80 years old,
* American Society of Anesthesiologists Physical Status (ASA-PS) risk groups of 1 to 3
* Elective thoracic surgery
* Operational types of thoracic surgery include; either open lung resection with thoracotomy or video-assisted thoracic surgery (VATS) operative procedure along with general a anesthesia, DLT insertion, and OLV for all patients

Exclusion Criteria:

* Refusal to participate in a study,
* History of severe asthma,
* Severe renal and hepatic insufficiencies,
* Pregnancy,
* History of previous pulmonary resection,
* Hemoglobinopathies.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From a total of fifty-nine patients, 50 patients underwent either video-assisted thoracic surgery or open thoracotomy after a diagnosis of a suspicious lung tumor.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Main Outcome Measure-(1) | Baseline time point after patient's arrival into operating room before anesthesia induction during elective thoracic operation
  Baseline time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(2) | Preoxygenation time point before anesthesia induction during elective thoracic operation
  Preoxygenatiom time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(3) | Third time point during thoracic operation defined as; five minutes after tracheal intubation during two-lung ventilation in the supine position during elective thoracic operation
  Third time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(4) | Fourth time point during thoracic operation defined as; 5 minutes after placing the patient in a lateral position with two-lung ventilation during elective thoracic operation
  Fourth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(5) | Fifth time point during thoracic operation defined as; at 1 minute after OLV placement during elective thoracic operation
  Fifth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(6) | Sixth time point during thoracic operation defined as; at 2 minute after OLV placement during elective thoracic operation.
  Sixth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(7) | Seventh time point during thoracic operation defined as; at 5 minute after OLV placement during elective thoracic operation.
  Seventh time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(8) | Eighth time point during thoracic operation defined as; at 10 minute after OLV placement during elective thoracic operation.
  Eighth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(9) | Ninth time point during thoracic operation defined as; at 15 minute after OLV placement during elective thoracic operation.
  Ninth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(10) | Tenth time point during thoracic operation defined as; at 30 minute after OLV placement during elective thoracic operation.
  Tenth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(11) | Eleventh time point during thoracic operation defined as; at 45 minute after OLV placement during elective thoracic operation.
  Eleventh time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(12) | Twelfth time point during thoracic operation defined as; at 60 minute after OLV placement during elective thoracic operation.
  Twelfth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation
Main Outcome Measure-(13) | Thirteenth time point during thoracic operation defined as; at 90 minute after OLV placement during elective thoracic operation.
  Thirteenth time point measurement of oxygen reserve index (ORi) equals to zero for predicting hypoxemia during one-lung ventilation

SECONDARY OUTCOMES:
Secondary Outcome-(1) | During anesthesia induction and maintenance of elective thoracic operation
  A correlation between ORi and peripheral oxygen saturation (SpO2), ORi and perfusion index (PI), and ORi pleth variability index (PVI) parameters that we collected during operation in patients undergoing elective thoracic surgery and one-lung ventilation (OLV)
Secondary Outcome-(2) | Twenty-four hours prior to elective thoracic surgery operation
  The Patients' demographic parameters and co-morbid diseases
Secondary Outcome-(3) | During elective thoracic surgery every five minutes continuously
  Measurement of mean arterial pressure (MAP)
Secondary Outcome-(4) | During elective thoracic surgery every five minutes continuously
  Measurement of systolic blood pressure (SBP)
Secondary Outcome-(5) | During elective thoracic surgery every five minutes continuously
  Measurement of diastolic blood pressure (DBP)
Secondary Outcome-(6) | During elective thoracic surgery every five minutes continuously
  Measurement of heart rate (HR)
Secondary Outcome-(7) | Five minutes after placing the patient in a lateral position with two-lung ventilation
  Arterial blood gas analysis during elective thoracic surgical operation

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Umit, MD, Study Chair — Trakya University, Trakya University Training and Research Hospital, Edirne, Turkey, 22030
Locations (1):
- Trakya University Training and Research Hospital, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Our data and statistical analysis of each investigated all parameter and data are available after the publication of the clinical study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available after the publication of our data upon request from the researchers.
Access Criteria: There is no internet website to obtain data but the researchers can contact Dr. Gonul Sagiroglu or Dr. Ayse Baysal.

REFERENCES:
- [Background] Karzai W, Schwarzkopf K. Hypoxemia during one-lung ventilation: prediction, prevention, and treatment. Anesthesiology. 2009 Jun;110(6):1402-11. doi: 10.1097/ALN.0b013e31819fb15d. PMID 19417615
- [Background] Applegate RL 2nd, Dorotta IL, Wells B, Juma D, Applegate PM. The Relationship Between Oxygen Reserve Index and Arterial Partial Pressure of Oxygen During Surgery. Anesth Analg. 2016 Sep;123(3):626-33. doi: 10.1213/ANE.0000000000001262. PMID 27007078
- [Result] Alday E, Nieves JM, Planas A. Oxygen Reserve Index Predicts Hypoxemia During One-Lung Ventilation: An Observational Diagnostic Study. J Cardiothorac Vasc Anesth. 2020 Feb;34(2):417-422. doi: 10.1053/j.jvca.2019.06.035. Epub 2019 Jun 28. PMID 31362907
- [Result] Chen ST, Min S. Oxygen reserve index, a new method of monitoring oxygenation status: what do we need to know? Chin Med J (Engl). 2020 Jan 20;133(2):229-234. doi: 10.1097/CM9.0000000000000625. PMID 31904726
- [Result] Campos JH, Sharma A. Predictors of Hypoxemia During One-Lung Ventilation in Thoracic Surgery: Is Oxygen Reserve Index (ORi) the Answer? J Cardiothorac Vasc Anesth. 2020 Feb;34(2):423-425. doi: 10.1053/j.jvca.2019.08.017. Epub 2019 Aug 18. No abstract available. PMID 31500971
- [Result] Koishi W, Kumagai M, Ogawa S, Hongo S, Suzuki K. Monitoring the Oxygen Reserve Index can contribute to the early detection of deterioration in blood oxygenation during one-lung ventilation. Minerva Anestesiol. 2018 Sep;84(9):1063-1069. doi: 10.23736/S0375-9393.18.12622-8. Epub 2018 May 14. PMID 29756744
- [Derived] Sagiroglu G, Baysal A, Karamustafaoglu YA. The use of oxygen reserve index in one-lung ventilation and its impact on peripheral oxygen saturation, perfusion index and, pleth variability index. BMC Anesthesiol. 2021 Dec 20;21(1):319. doi: 10.1186/s12871-021-01539-8. PMID 34930139